CLINICAL TRIAL: NCT01976208
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled Clinical Study to Evaluate the Safety and Efficacy of Recombinant Humanized Anti-IgE Monoclonal Antibody Injection(Omalizumab) in Patients With Allergic Asthma
Brief Title: Safety and Efficacy Study of Omalizumab to Treat Allergic Asthma
Acronym: AA007
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Zhangjiang Biotechnology Limited Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMAB007
Record Dates: First submitted 2013-10-23; First posted 2013-11-05 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Allergic Asthma
Keywords: Omalizumab; IgE; Asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omalizumab (Experimental): During the 4~6-week Run-in phase, the dosage of budesonide inhaled powder(BUD) was prescribed and optimized to maintain asthma control according to Global Initiative for Asthma(GINA, 2008) guidelines. During the following treatment phase, patients continued to receive optimized BUD and Omalizumab for 28 weeks, administered by subcutaneous injection every 2 weeks or 4 weeks. The dosage of Omalizumab received was based on body weight and serum IgE.
  Interventions: Drug: Omalizumab
- placebo (Placebo Comparator): During the 4~6-week Run-in phase, the dosage of budesonide inhaled powder(BUD) was prescribed and optimized to maintain asthma control according to Global Initiative for Asthma(GINA, 2008) guidelines. During the treatment phase, patients continued to receive placebo and optimized BUD for 28 weeks, administered by subcutaneous injection every 2 weeks or 4 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Omalizumab — The recommended dose is 0.016mg/kg/IgE(IU/ml) every 4 weeks. It is administered by subcutaneous injection.If the total dose per 4 weeks is 150~300mg, the dosing interval will be every 4 weeks; if the total dose per 4 weeks is 450mg~750mg，then dosing interval is every 2 weeks.
  Other Names: other name: Aomaishu; Recombinant Humanized Anti-IgE Monoclonal Antibody
  Arms: Omalizumab
Drug: placebo
  Arms: placebo

SUMMARY:
The primary purpose is to evaluate the safety and efficacy of recombinant humanized anti-IgE monoclonal antibody injection in patients with allergic asthma.

DETAILED DESCRIPTION:
Omalizumab will be given as add-on treatment to budesonide inhaled powder in patients with moderate or severe allergic asthma(IgE>=60IU/ml), who demonstrate inadequate asthma symptom control. Response to Omalizumab will be assessed by the overall improvement in control of asthma.

Omalizumab is a recombinant humanized monoclonal antibody that selectively binds to human immunoglobulin E(IgE). The antibody has a molecular weight of approximately 150 kilodaltons and produced by Chinese Hamster Ovary cell.

Omalizumab inhibits the binding of IgE to the high-affinity IgE receptor on the surface of mast cells and basophils. Reduction in surface-bound IgE on cells limits the degree of release of mediators of the allergic response.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 15~65 years
* Written informed consent provided
* Total serum IgE >=60IU/ml
* Duration of allergic asthma >= 1 year according to GINA(2008)
* Poor response to moderate to high dose inhaled corticosteroid (400ug/day~800ug/day) >= 4 weeks
* Agreed to be not pregnant, contraception during study and later 6 months.

Exclusion Criteria:

Patients who met the below criteria were excluded:

* Be regular smokers(>10 cigarettes per day and for at least 2 years)
* Patients who are currently pregnant or nursing or intend to become pregnant over the course of the study or later 6 months
* COPD, according to the guideline of Chinese society of respiratory diseases
* An active lung disease other than allergic asthma
* Patients with significant underlying medical conditions
* Allergic to immunoglobin or any formulation ingredient of the product
* Patients with diabetes or uncontrolled hypertension(Systolic blood pressure>160mmHg or Diastolic blood pressure>95mmHg)
* HIV positivity or cancer patient
* Prior exposure to Xolair

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2010-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with asthma exacerbation | 32 weeks

SECONDARY OUTCOMES:
Pulmonary function measured by FEV1 and FEV1/FVC | 32 weeks
Asthma symptoms evaluated by patients by using the Questionaire, Asthma Quality of Life Questionaire | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nanshan Zhong, M.D., Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (27):
- China (27):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - The Second Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Chongqing Xinqiao Hospital, Chongqing
  - Chinese PLA Fuzhou General Hospital of Nanjing Military Command, Fuzhou
  - South Hospital of South Medical University, Guangzhou
  - Sir Run Run Shaw Hospital of Zhejiang University, Hangzhou
  - The First Affiliated Hospital of Zhejiang University, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou
  - Chinese PLA Jinan Military General Hospital, Jinan
  - Shandong Provincial Hospital, Jinan
  - Jiangsu Province Hospital, Nanjing
  - Zhongda Hospital, Southeast University, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Qingdao Municipal Hospital, Qingdao
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai
  - Chinese PLA Shenyang Military Command General Hospital, Shenyang
  - The First hospital of China Medical University, Shenyang
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - The Second Hospital of Tianjin Medica University, Tianjin
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and technology, Wuhan
  - Xi'an Xijing Hospital, Xi'an